CLINICAL TRIAL: NCT04229641
Title: Fall Prevalence and Factors Affecting Falls in Elderly.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Emine Handan Tüzün, Professor, Eastern Mediterranean University
Other Study IDs: ETK00-2019-0175
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Falling

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Falling in the elderly is a common problem that can have devastating consequences for individuals and affect social support networks. Falls are considered to be the most common cause of injury in the elderly population. In developed countries, it is reported that one out of every three elderly people in the society has fallen during the year and that number has increased gradually after the age of 65. There are many risk factors that cause falls in the elderly. These factors may be caused by the elderly itself (intrinsic) or the environment (extrinsic).

The aim of this study are two folds:

1. To determine the prevalence of falls in the last year among the elderly living in Degirmenlik region of Nicosia, Northern Cyprus,
2. To determine predictors of the risk of falls in the elderly.

DETAILED DESCRIPTION:
Falling in the elderly is a common problem that can have devastating consequences for individuals and affect social support networks. Falls are considered to be the most common cause of injury in the elderly population. In developed countries, it is reported that one out of every three elderly people in the society has fallen during the year and that number has increased gradually after the age of 65. As a result of the falls, significant burdens on health services are imposed. In this context, determining the risk factors that cause falls is as important as public health as well as preventive physiotherapy services.There are many risk factors that cause falls in the elderly. These factors may be caused by the elderly itself (intrinsic) or the environment (extrinsic). Most of falls are caused by interactions between multiple risk factors. However, in individuals aged 75 years and over, even 10% of those without risk factors have been reported to fall at any time during the year.However, all these factors may vary from country to country depending on the cultural differences and living conditions of the elderly.

Therefore, it is important to investigate the risk factors that cause falls in each population to prevent falls.

The aim of this study are two folds:

1. to determine the prevalence of falls in the last year among the elderly living in Degirmenlik region of Nicosia, Northern Cyprus,
2. To determine predictors of the risk of falls in the elderly.

The population of the cross-sectional study consists of 1486 people aged 65 years and over living in 16 villages of Degirmenlik Municipality of Nicosia, Northern Cyprus.

The following formulas were used to determine the sample size.

n= z² x p(1-p) ̸ Є²

n'= n ̸ 1+ (z² x p (1-p) ̸ Є² N

(z = z score; ɛ = %95 margin of error in confidence interval; N= universe size ve p = prevalence) First sample size z = 1,96; with assumptions ɛ = 0,05 and p = 0.50 it was calculated as 384 people. The final sample size was calculated as 499 people, with a non-response rate of 30%. In this context, 499 elderly individuals selected by simple random sampling method will form the sample of the study.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older,
* Residing in one of the villages of Degirmenlik Municipality
* To be able to walk independently or with walking aid.

Exclusion Criteria:

* People who cannot cooperate
* People with acute illnesses

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The population of the study consists of 1486 people aged 65 years and over living in 16 villages of Degirmenlik Municipality.
Sampling Method: Probability Sample
Enrollment: 499 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
prevalence | last one year period
  fall prevalence

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Hacıküçük, BSc., PT., Principal Investigator — Eastern Mediterranean University
Locations (1):
- 1. Eastern Mediterranean University Health Sciences Faculty, Department of Physiotherapy and Rehabilitation,, Mersin, Northern Cyprus, Turkey (Türkiye)